CLINICAL TRIAL: NCT01306474
Title: Clinical Study on the Regulatory T Cells in the Uveitis Patients Treated by Methotrexate
Brief Title: Observation on the Treg in the Uveitis Patients
Acronym: OTUP
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: licai/the eye department of xijing hospital
Other Study IDs: xjyy090706
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Uveitis
Keywords: CD4/CD25 Tr cell,TNF,IFN-γ,IL-2
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Experimental:A Drug: prednisone profess to convinced 1-1.5mg/Kg.d Experimental:B Drug: methotrexate profess to convinced 7.5-15mg/w, concoction prednisone profess to convinced 0.5-1mg/Kg.d
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prednisone: profess to convinced 1-1.5mg/Kg.d
- methotrexate to band prednisone: profess to convinced 7.5-15mg/w, concoction prednisone profess to convinced 0.5-1mg/Kg.d

SUMMARY:
AIM: To study the expression of CD4+CD25+ high regulatory T cells in peripheral blood of patients with uveitis and to explore its role in the development of uveitis.

DETAILED DESCRIPTION:
Uveitis describes inflammation that exists in the uveal tract, but the disease course has such a variety of manifestations. Uveitis (intraocular inflammatory diseases) includes sight-threatening diseases such as Behcet disease, birdshot retinochoroidopathy, Vogt-Koyanagi-Harada, sympathetic ophthalmia and ocular sarcoidosis, and may be of infectious or autoimmune etiology.

CD4+ CD25+ Tr cells play a key role in the maintenance of peripheral self-tolerance by inhibiting the activation and proliferation of unreactive T cells. In addition to a direct suppressor effect on CD4+CD25+ Tr cells. CD4+CD25+ Tr cells may regulate the immune response through dendritic cell. Like cytotoxic T-lymphocytes and natural killer cells,activated human CD4+CD25+ Tr cells display perforin-dependent cytoxicity against autologous target cell, including activated CD4+ and CD8+ T cells.

Experimental autoimmune uveoretinitis (EAU) is a model of uveitis. Regulatory T cells in the uveitis are currently thought to be the etiologic agent of uveitis because IFN-γ,IL-2(interleukin-2),TNF(Tumor Necrosis Factor alpha) levels are elevated in the retina during uveitis Following stimulation with IL-2 expression was upregulated in PBMC(peripheral blood mononuclear cell) of healthy subjects and patients with scleritis or uveitis. By ELISA, we confirmed that IL-2 induced the secretion of the protein in human PBMC and in mouse CD4+T cells. Experiment found, by an intracellular cytokine analysis assay, that the IFN-γ,IL-2,TNF expressing cells were predominantly CD4+T cells with a memory phenotype. Consistent with our RNA data, the percentage of CD4+T cells was higher in scleritis patients than in healthy subjects.

We analyzed peripheral blood of thirty uveitis patients enrolled in Department of Ophthalmology, Xijing Hospital clinical trials. The demographics of the patients, including age, sex, diagnosis and medications at time of sample collection .

Biospecimen Description:

Experimental: A Drug: prednisone profess to convinced 1-1.5mg/Kg.d Experimental: B Drug: methotrexate profess to convinced 7.5-15mg/w, concoction prednisone profess to convinced 0.5-1mg/Kg.d Methods CD4+CD25+ Tr cells, CTLA-4 and an intracellular cytokine analysis assay that the IFN-γ,IL-2,TNF expressing cells were measured in 30 uveitis patients before and after 1 month,3 months of prednisone and methotrexate.

Cytokine assays. For intracellular cytokine detect, CD4+T cells were cultured as indicated above and restimulated for 5h with 1mg/ml phorbol 12-myristate 13-acetate (PMA) and ionomycin (1mg/ml) in the presence of Golgistop, we added antibodies (IFN-γ,IL-2,TNF). We performed cytokine staining using BD Biosciences and analyzed samples by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 60 years
* the first episode

Exclusion Criteria:

* had other intracranial pathologies (e.g.tumor,infection)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ages eligible for Study:18 Years to 60 Years. Study Population had two eye attacks in a year.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: li cai, MD, Study Chair — the ophthalmology department, xijing Hospital
Locations (1):
- Department of Ophthalmology, Xijing Hosptial, Xi'an, Shaanxi, China